CLINICAL TRIAL: NCT01290484
Title: An Investigational Pilot Study to Evaluate Sildenafil for the Treatment of Lymphatic Malformations
Brief Title: A Study to Evaluate Sildenafil for the Treatment of Lymphatic Malformations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alfred Lane, Professor of Dermatology and of Pediatrics, Emeritus, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-10202010-7129; UL1TR000093 (NIH)
Record Dates: First submitted 2011-02-03; First posted 2011-02-07 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-05

CONDITIONS: Lymphangioma
Keywords: Lymphatic malformation, vascular malformation
MeSH Terms: conditions — Lymphangioma; Lymphatic Abnormalities; Vascular Malformations | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental): Sildenafil oral tablet three times daily
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Sildenafil oral tablet three times daily
  Other Names: Revatio; Viagra

SUMMARY:
There is an unsatisfied medical need for a first-line treatment of lymphatic malformations with a good benefit/risk profile. Based on a patient experience in the institution, the investigators plan to verify whether or not the medication sildenafil has a beneficial effect on lymphatic malformations. The investigators plan to do this by treating patients with lymphatic malformations with the medication sildenafil for a 20 week period. This is an investigator initiated study funded by an Innovations in Patient Care grant and a SPARK grant.

DETAILED DESCRIPTION:
Lymphatic malformations can be challenging to treat. Mainstay interventions including surgery and sclerotherapy are invasive and can result in local recurrence and complications. We sought to assess the effect of 20 weeks of oral sildenafil on reducing lymphatic malformation volume and symptoms in children. Seven children (4 boys, 3 girls; ages 13-85 months) with lymphatic malformations were given oral sildenafil for 20 weeks in this open-label study. The volume of the lymphatic malformation was calculated blindly using magnetic resonance imaging performed before and after 20 weeks of sildenafil. Lymphatic malformations were assessed clinically on weeks 4, 12, 20, and 32. Both the physician and parents evaluated the lymphatic malformation in comparison with baseline. Sildenafil can reduce lymphatic malformation volume and symptoms in some children. ( J Am Acad Dermatol 2014;70:1050-7.)

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent(s) for study participation and (where applicable) the use of the participant's images are obtained according to national regulations from the participant's parent(s) or guardian(s) prior to performing any study procedures.
2. The participant is 6 months to 10 years of age at inclusion.
3. The participant weight is at least 8kg.
4. A diagnosis of LM or mixed venous lymphatic malformation involving the skin and subcutaneous tissue and at least 3cm based on clinical and radiographic criteria.
5. LMs may benefit from systemic therapy based on clinical criteria.
6. Females must not be pregnant or breast-feeding.
7. If participant is a child, parent/guardian must be able to follow instructions and must be willing and able to ensure that the subject is present for all required study visits.
8. Subject has no contraindication for use of sildenafil.
9. LMs may involve any part of the body.
10. Subject will have normal results on screening tests (eye exam, blood tests).
11. Subject has no contraindication for MRI examinations, such as metal implants, etc.
12. Subject must not be a smoker.

Exclusion Criteria:

1. The participant has a medically unstable health status that may interfere with his/her ability to complete the study.
2. The participant presents with one or more of the following medical conditions: hepatic impairment; severe renal impairment; lymphedema conditions such as Milroy disease, Meige lymphedema, Hennekam syndrome, Njolstad syndrome, Aagenaes syndrome, and Fabry disease; hypotension or at risk for hypotension; seizures or history of seizures; any significant cardiovascular risk factors and any condition which requires participants to use nitric oxide donors or nitrates in any form; underlying anatomic or vascular risk factors for developing non-arteritic anterior ischemic optic neuropathy (NAION) including low ocular cup to disc ratio, age over 10, diabetes, hypertension, coronary artery disease, hyperlipidemia, and smoking. (Participants with Down syndrome, Turner syndrome, and Noonan syndrome will be considered on a case-by-case basis).
3. The participant has received at least one of the following medications contraindicated in association with sildenafil within 15 days of inclusion: Alprostadil, Azole antifungals, Clarithromycins, Conivaptan, Delavirdine, Erythromycins, Fluvoxamine, Grapefruit, Imatinib, Nefazodone, Nitrates/sodium thiosulfate, Non-selective and selective alpha blockers, Protease inhibitors, Rufinamide, Tadalafil, Telithromycin, Vardenafil, Yohimbe, Yohimbine, Amifostine, Lapatinib, Warfarin
4. The participant requires concomitant use of potent cytochrome P450 3A4 inhibitors (such as ketoconazole, itraconazole, erythromycin, saquinavir) or concomitant use of ritonavir.
5. The patient has had extensive prior surgery or sclerotherapy to treat LM such that scarring may interfere with the treatment effect of sildenafil.
6. The participant has previously been administered treatment for LMs or surgical procedures have been performed to remove the index LMs.
7. Participant is currently pregnant or considering becoming pregnant in the next 20 weeks.
8. The participant is known to have an allergy to sildenafil.
9. Ulcerated or currently infected LMs with pain.
10. Diagnosis of the soft tissue tumor as LM is not clinically certain.
11. The participant is participating in another clinical study.
12. The participant has a history of priapism or is diagnosed with sickle cell anemia or any other disorder which may predispose to priapism.
13. The investigator may declare any subject ineligible for a valid medical reason.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred T Lane, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Danial C, Tichy AL, Tariq U, Swetman GL, Khuu P, Leung TH, Benjamin L, Teng J, Vasanawala SS, Lane AT. An open-label study to evaluate sildenafil for the treatment of lymphatic malformations. J Am Acad Dermatol. 2014 Jun;70(6):1050-7. doi: 10.1016/j.jaad.2014.02.005. Epub 2014 Mar 20. PMID 24656411

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: Participants were given sildenafil for 20 weeks. Participants weighing more than 20 kg were given 20 mg 3 times daily (60 mg/day). Participants weighing between 8 kg and 20 kg were given 10 mg 3 times daily (30 mg/day).
Period: Overall Study
Arm/Group | Sildenafil
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Based on funding
Groups:
- Sildenafil: Male and female subjects between the ages of 6 months and 10 years, weighing at least 8 kg and had been given a diagnosis of a lymphatic malformation of at least 3 cm based on clinical and radiologic criteria. Macrocystic, microcystic, or mixed lymphatic malformations involving any location on the body were included. Lymphatic malformations associated with an incomplete response to previous treatments, a risk of functional or aesthetic impairment, or local complications were included.
Arm/Group | Sildenafil
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: months] | 51.3 [13 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7
Weight [Mean (Full Range); unit: Kilograms] | 17.0 [9.7 to 24.2]

OUTCOME MEASURES:

1. Primary Outcome: Change in Volume of Lymphatic Malformation
Description: Participants were given sildenafil for 20 weeks. Participants weighing more than 20 kg were given 20 mg 3 times daily (60 mg/day). Participants weighing between 8 kg and 20 kg were given 10 mg 3 times daily (30 mg/day).
Time Frame: Baseline, 20 weeks
Measure: Number; unit: percentage of volume change
Groups:
- Sildenafil: The primary outcome was the effect of sildenafil on lymphatic malformation volume. Response to sildenafil was characterized by any decrease in lymphatic malformation volume. Lymphatic malformations volumes were assessed blindly by MRI volume segmentation analysis at baseline and after 20 weeks of sildenafil. 4 subjects had a lymphatic malformation volume decrease.
Arm/Group | Sildenafil
Number analyzed (Participants) | 7
percentage of volume change
  Subject 1 | 3.7
  Subject 2 | -4.3
  Subject 3 | -1.0
  Subject 4 | -31.7
  Subject 5 | -21.7
  Subject 6 | 1.1
  Subject 7 | 29.6
Statistical Analysis 1: Comparison: Sildenafil; Test type: Superiority or Other; Mean percentage volume change = -3.47

ADVERSE EVENTS:
Time Frame: 20 weeks on sildenafil and 12 weeks after sildenafil
Description: Participants were given sildenafil for 20 weeks. Participants weighing more than 20 kg were given 20 mg 3 times daily (60 mg/day). Participants weighing between 8 kg and 20 kg were given 10 mg 3 times daily (30 mg/day).
Groups:
- Sildenafil: Adverse events reported while one sildenafil were minimal. All subjects tolerated the prescribed medication dose. One subject developed an upper respiratory tract infection and experienced temporary hearing loss due to fluid accumulation. This was resolved completely and she experienced no further hearing loss while on sildenafil. Four parents requested to have the child continue sildenafil after study completion.
Arm/Group | Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil (N=7)
Nausea/indigestion (Gastrointestinal disorders) | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Mild insomnia (Psychiatric disorders) | 3
Fever (Investigations) | 2
Emesis (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 1
Epistaxis (Blood and lymphatic system disorders) | 1
Prolonged erections (Reproductive system and breast disorders) | 1
Temporary hearing illness (Infections and infestations) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Bleeding into lymphangioma circumscriptum (Blood and lymphatic system disorders) | 1

LIMITATIONS AND CAVEATS:
Baseline MRI examinations were performed within 6 months prior to commencement of sildenafil; several subjects took sildenafil for more than 20 weeks due to MRI scheduling and personal accommodations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No